CLINICAL TRIAL: NCT02534428
Title: The Effects of Superfine Merino Wool in the Management of Childhood Atopic Dermatitis
Brief Title: Wool Clothing for the Management of Childhood Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Australian Wool Innovation Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 34037 A
Record Dates: First submitted 2015-08-11; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- wool-first (wool-standard) (Experimental): superfine merino wool clothing to be worn for 6 weeks followed by 6 weeks of standard clothing (cotton)
  Interventions: Other: wool clothing
- cotton-first (standard-wool) (Active Comparator): standard (cotton) clothing to be work for 6 weeks followed by 6 weeks of superfine merino wool clothing
  Interventions: Other: wool clothing

INTERVENTIONS:
Other: wool clothing — superfine merino wool ensembles for baby wear

SUMMARY:
The study is a sequentially recruited, cross-over-cohort, outpatient-based evaluation of the effectiveness of wool clothing, as compared to standard clothing, in reducing the severity of childhood atopic dermatitis over two consecutive six-week periods.

DETAILED DESCRIPTION:
The study will aim for a sample size of approximately 40 patients between the ages of 0 and 3 years of children referred to the Dermatology Department at the Royal Children's Hospital for management of mild to moderate atopic dermatitis. They will be sequentially recruited and randomized to the wool-standard clothing arm or standard clothing-wool arm.

The study will run for 12 weeks for each participant with two 6-week periods, either of wool followed by standard clothing or standard followed by wool clothing. Participants will be assessed by a blinded trained researcher during this time, at their initial appointment, 3 weeks, 6 weeks, 9 weeks and 12 weeks.

The primary outcome is change in the severity of atopic eczema at 6 weeks. Severity of atopic eczema will be measured using the Scoring Atopic Dermatitis (SCORAD) index.

Secondary outcomes include the change in the severity of eczema using the SCORAD at 3 weeks and the Atopic Dermatitis Severity Index (ADSI) score at 3 and 6 weeks and quality of life assessment using the Dermatology Life Quality Index (DLQI) at 3 and 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate eczema as determined by a SCORAD of 1-50 at their initial visit
* has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participants behalf
* is capable of returning for review having had education through the Royal Children's Hospital eczema workshop

Exclusion Criteria:

* known reactions to wool products
* is unable to attend visits
* has unstable eczema defined by treatment escalation or increased topical anti-inflammatory use in the preceding 2 months

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in the SCORAD Scoring Atopic Dermatitis Index (Units on a scale) | at 6 weeks
  blinded assessor administered SCORAD

SECONDARY OUTCOMES:
Change in the SCORAD Scoring Atopic Dermatitis Index (Units on a scale) | at 3 weeks
  blinded assessor administered SCORAD
Change in ADSI Atopic Dermatitis Severity Index (Units on a scale) | at 6 weeks
  blinded assessor administered ADSI
Change in ADSI Atopic Dermatitis Severity Index (Units on a scale) | at 3 weeks
  blinded assessor administered ADSI
Change in IDQOL Infant's Dermatitis Quality of Life index (Units on a scale) | at 6 weeks
Change in IDQOL Infant's Dermatitis Quality of Life index (Units on a scale) | at 3 weeks

OTHER OUTCOMES:
change in moisturiser use (times per day) | at 6 weeks
change in moisturiser use (times per day) | at 3 weeks
change in topical steroid use (times per day) | at 6 weeks
change in topical steroid use (times per day) | at 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John C Su, FRACP FACD, Principal Investigator — Murdoch Childrens Research Institute

REFERENCES:
- [Background] Ricci G, Patrizi A, Bellini F, Medri M. Use of textiles in atopic dermatitis: care of atopic dermatitis. Curr Probl Dermatol. 2006;33:127-43. doi: 10.1159/000093940. PMID 16766885
- [Background] Mason R. Fabrics for atopic dermatitis. J Fam Health Care. 2008;18(2):63-5. PMID 18512638
- [Background] Hatch KL, Maibach HI. Textile fiber dermatitis. Contact Dermatitis. 1985 Jan;12(1):1-11. doi: 10.1111/j.1600-0536.1985.tb01030.x. PMID 3884253
- [Background] Gelmetti C, Wollenberg A. Atopic dermatitis - all you can do from the outside. Br J Dermatol. 2014 Jul;170 Suppl 1:19-24. doi: 10.1111/bjd.12957. Epub 2014 May 9. PMID 24720530
- [Result] Bendsoe N, Bjornberg A, Asnes H. Itching from wool fibres in atopic dermatitis. Contact Dermatitis. 1987 Jul;17(1):21-2. doi: 10.1111/j.1600-0536.1987.tb02638.x. PMID 3652686